CLINICAL TRIAL: NCT01693146
Title: Evaluation of Safety and Efficacy of Short-time TNI® Treatment in Patients With COPD and Hypercapnia Acute Testing of Oxygen Demand Using TNI® vs. Standard Insufflation in COPD Patients With Hypercapnia at Rest
Brief Title: STIT-2: Evaluation of Safety and Efficacy of Short-time TNI® Treatment in Patients With COPD and Hypercapnia
Acronym: STIT-2
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: TNI Medical AG (Industry)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. Christian M. Kaehler, a.Univ.-Prod. Dr., Medical University Innsbruck
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UN4484; UN4484 (Other: Ethic Committee Innsbruck)
Record Dates: First submitted 2012-09-14; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: COPD; Hypercapnia
Keywords: Oxygen; High Flow; COPD; Hypercapnia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal insufflation of oxygen (Active Comparator): Nasal insufflation of oxygen starting at at flow of 0.5 L/min.
  Interventions: Device: Nasal insufflation of oxygen
- Nasal oxygen insufflation with a TNI® 20 oxy device (Active Comparator): Device: TNI®20 oxy Nasal insufflation at a constant high flow of 15 L/min with oxygen addition starting at 0.5 L/min
  Interventions: Device: Nasal oxygen insufflation with a TNI® 20 oxy device

INTERVENTIONS:
Device: Nasal oxygen insufflation with a TNI® 20 oxy device — Nasal insufflation at a constant high flow of 15 L/min with oxygen addition starting at 0.5 L/min
  Arms: Nasal oxygen insufflation with a TNI® 20 oxy device
Device: Nasal insufflation of oxygen — Nasal insufflation of oxygen starting at at flow of 0.5 L/min.
  Arms: Nasal insufflation of oxygen

SUMMARY:
Evaluation of Safety and Efficacy of Short time TNI Treatment in Patients with COPD and hypercapnia.

Acute testing of oxygen demand using TNI vs. standard oxygen application in stable COPD patients with hypercapnia.

DETAILED DESCRIPTION:
TNI, the nasal insufflation of a high flow of warm, humidified air, is an extremely comfortable and uncomplicated alternative to numerous other approaches in non-invasive ventilation (NIV). Up to now, NIV therapy could only be applied by masks with the associated complications as patients could not tolerate high airflow delivered by a thin nasal cannula without humidification and warming, thus causing concomitant negative effects. The new therapy TNI shows a high rate of acceptance by children, too.

At present, there are two different types of devices available for nasal insufflation in clinics:

TNI 20s, an air humidifier for clinical compressed air, and the TNI20 oxy, an air humidifier for clinical compressed air, which can be combined with oxygen.

TNI 20 oxy The system, which is unique throughout the world, is optimized for the application of flows of up to 20L/min and fulfils the minimum requirements of the "American Society of Testing and Materials" for a high flow air humidifier in the non-invasive application of 10 mg H2O/L (equivalent to about 60% rel. humidity at an ambient temperature of 22°C) for the air humidity. The warming of the air flow by 5-15°C can be adjusted relative to the ambient temperature. Condensation is prevented in the nasal applicator by heating the tube as far as the nostrils. The device automatically controls humidity and temperature depending on the prevailing ambient conditions. The TNI®20s can be attached to the hospital infrastructure by means of a standard pressure regulator.

In another ongoing study (STIT-1) TNI 20 oxy was evaluated for its safety in COPD patients without hypercapnia. In a first interim analysis which included 14 patients high flow oxygen delivery was safe.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with an indication for long-term oxygen therapy (LTOT)
* Presence of hypercapnia at rest without oxygen supplementation (PaCO2 > 45 mmHg)
* Age 30 - 85 years
* Functional GOLD class: COPD GOLD IV as defined by the following:

FEV1/FVC < 70% and a Post-bronchodilator FEV1 < 30% or FEV1 < 50% and a PaO2 < 60 mmHg and/or PaCO2 > 50 mmHg

Exclusion Criteria:

* Clinical instability of the patient
* No lung function testing possible
* Exacerbation within the last 14 days prior to inclusion into the study
* Serious concomitant diseases that may jeopardize the inclusion of the patient into the study from the investigator's point of view
* Severe anaemia, defined by a haemoglobin <8.5 G/L
* Participation of the patient in any other ongoing study

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
PaO2 | 60 min
  Change in the partial oxygen pressure in the arterial blood (blood gas analysis) at a defined oxygen flow rate (L/min)

SECONDARY OUTCOMES:
O2% | 60 min
  Change in the oxygen saturation in the arterial blood (blood gas analysis) at a defined oxygen flow rate (L/min)
PaCO2 | 60 min
  Change in the PaCO2 in the arterial blood (blood gas analysis) at a defined oxygen flow rate (L/min)
AaDO2 | 60 min
  Change in the AaDO2 in the peripheral blood at a defined oxygen flow rate (L/min)
RV and TLC | 60 min
  No increase in the residual volume (RV) and the total lung capacity (TLC) > 15% of the mean actual value at visits 1 and 2 (measurement 60 + 10 minutes after oxygen insufflation with a TNI system).

CONTACTS AND LOCATIONS:
Overall Officials: Christian M Kaehler, MD, Principal Investigator — Medical University Innsbruck
Locations (4):
- Christian Kähler, Innsbruck, Austria
- Germany (2):
  - Pneumologie, Medizinische Klinik und Poliklinik I, University of Dresden, Dresden
  - Klinik für Innere Medizin V, Universitätsklinikum Homburg, University of Homburg/Saar, Homburg
- Klinik und Poliklinik für Pneumologie, Inselspital Berne, University of Berne, Bern, Switzerland

REFERENCES:
- [Derived] Vogelsinger H, Halank M, Braun S, Wilkens H, Geiser T, Ott S, Stucki A, Kaehler CM. Efficacy and safety of nasal high-flow oxygen in COPD patients. BMC Pulm Med. 2017 Nov 17;17(1):143. doi: 10.1186/s12890-017-0486-3. PMID 29149867